CLINICAL TRIAL: NCT06327750
Title: The Microcirculation, Dialysis Modality and Sequestered Salt
Acronym: MIMOSA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Dutch Kidney Foundation (Other); Niercentrum aan de Amstel (Unknown); B.Braun Avitum AG (Industry)
Responsible Party: Principal Investigator, Muriel P.C. Grooteman, Principal Investigator, Internist-Nephrologist, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL83566.018.24
Record Dates: First submitted 2024-02-21; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: End-stage Renal Disease
Keywords: Hemodialysis; Hemodiafiltration; Microcirculation; Sequestered salt content
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Renal Dialysis

STUDY DESIGN:
Intervention Model Description: Randomized cross-over trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Hemodialysis (DNa=PNa) (Active Comparator): High-flux hemodialysis with expected diffusive zero sodium balance (DNa=PNa)
  Interventions: Device: Hemodialysis (DNa<PNa); Device: Hemodialysis after isolated ultrafiltration (DNa=PNa); Device: High volume hemodiafiltration (DNa=PNa); Device: High volume hemodiafiltration (DNa<PNa)
- Hemodialysis (DNa<PNa) (Active Comparator): High-flux hemodialysis with expected diffusive sodium efflux (DNa<PNa, difference: 3 mmol/L)
  Interventions: Device: Hemodialysis (DNa = PNa); Device: Hemodialysis after isolated ultrafiltration (DNa=PNa); Device: High volume hemodiafiltration (DNa=PNa); Device: High volume hemodiafiltration (DNa<PNa)
- Hemodialysis after isolated ultrafiltration (DNa=PNa) (Active Comparator): High-flux hemodialysis after isolated ultrafiltration with expected zero sodium balance (DNa=PNa)
  Interventions: Device: Hemodialysis (DNa = PNa); Device: Hemodialysis (DNa<PNa); Device: High volume hemodiafiltration (DNa=PNa); Device: High volume hemodiafiltration (DNa<PNa)
- High volume hemodiafiltration (DNa=PNa) (Active Comparator): High volume hemodiafiltration with expected diffusive zero sodium balance (DNa=PNa)
  Interventions: Device: Hemodialysis (DNa = PNa); Device: Hemodialysis (DNa<PNa); Device: Hemodialysis after isolated ultrafiltration (DNa=PNa); Device: High volume hemodiafiltration (DNa<PNa)
- High volume hemodiafiltration (DNa<PNa) (Active Comparator): High volume hemodiafiltration with expected diffusive sodium efflux (DNa<PNa, difference: 3 mmol/L)
  Interventions: Device: Hemodialysis (DNa = PNa); Device: Hemodialysis (DNa<PNa); Device: Hemodialysis after isolated ultrafiltration (DNa=PNa); Device: High volume hemodiafiltration (DNa=PNa)

INTERVENTIONS:
Device: Hemodialysis (DNa = PNa) — High-flux hemodialysis with an expected zero diffusive sodium balance (DNa = PNa)
  Arms: Hemodialysis (DNa<PNa); Hemodialysis after isolated ultrafiltration (DNa=PNa); High volume hemodiafiltration (DNa<PNa); High volume hemodiafiltration (DNa=PNa)
Device: Hemodialysis (DNa<PNa) — High-flux hemodialysis with expected diffusive sodium efflux (DNa<PNa, difference: 3 mmol/L)
  Arms: Hemodialysis (DNa=PNa); Hemodialysis after isolated ultrafiltration (DNa=PNa); High volume hemodiafiltration (DNa<PNa); High volume hemodiafiltration (DNa=PNa)
Device: Hemodialysis after isolated ultrafiltration (DNa=PNa) — High-flux hemodialysis after isolated ultrafiltration with an expected zero diffusive sodium balance (DNa=PNa)
  Arms: Hemodialysis (DNa<PNa); Hemodialysis (DNa=PNa); High volume hemodiafiltration (DNa<PNa); High volume hemodiafiltration (DNa=PNa)
Device: High volume hemodiafiltration (DNa=PNa) — High volume hemodiafiltration with an expected zero diffusive sodium balance (DNa=PNa) Convection volume: ≥23L/session
  Arms: Hemodialysis (DNa<PNa); Hemodialysis (DNa=PNa); Hemodialysis after isolated ultrafiltration (DNa=PNa); High volume hemodiafiltration (DNa<PNa)
Device: High volume hemodiafiltration (DNa<PNa) — High volume hemodiafiltration with expected diffusive sodium efflux (DNa<PNa, difference: 3 mmol/L) Convection volume: ≥23L/session
  Arms: Hemodialysis (DNa<PNa); Hemodialysis (DNa=PNa); Hemodialysis after isolated ultrafiltration (DNa=PNa); High volume hemodiafiltration (DNa=PNa)

SUMMARY:
The aim of this clinical trial is to investigate the effect of 5 different dialysis treatments (combinations of dialysis mode and dialysis fluid sodium content) on the microcirculation (MC) and sequestered sodium content (SSC) in adult prevalent end-stage kidney disease (ESKD) patients treated with hemodialysis (HD) or hemodiafiltration (HDF). The main questions it aims to answer are:

1. What are the effects on the sequestered sodium content and microcirculation after 4 weeks of treatment with the following dialysis modes?

   * HDF with an expected zero diffusive sodium balance (Dialysate sodium concentration (DNa)= Plasma sodium concentration (PNa)) compared to
   * HDF with an expected diffusive sodium efflux (DNa < PNa, difference 3 mmol/L) compared to
   * HD with an expected zero diffusive sodium balance (DNa = PNa) compared to
   * HD with an expected diffusive sodium efflux (DNa < PNa, difference 3 mmol/L) compared to
   * Isolated ultrafiltration for 30 minutes followed by HD with an expected zero diffusive sodium balance (DNa = PNa)
2. Are the SSC and MC interrelated in this patient group?

This study is a randomized cross-over trial. Participants will be subjected to the abovementioned dialysis treatment modes in random order.

DETAILED DESCRIPTION:
The life expectancy of patients with end-stage kidney disease (ESKD) is poor. Post-dilution online hemodiafiltration (HDF) is associated with a lower mortality than standard hemodialysis (HD), especially when a high convection volume is achieved (high-volume HDF; hvHDF). It is unclear, however, why (hv)HDF improves survival. Neither an increased clearance of middle molecular weight uremic toxins, nor an improved bio-incompatibility can explain the difference. As the effects are already observed within 2.5 years, recovery of a functional disorder is more likely than restoration of structural alterations. The recuperation of vascular dysfunction may be the missing piece of the puzzle. Previous literature showed (1) that the microcirculation (MC) is severely disturbed in dialysis patients, (2) excess sodium can bind to glycosaminoglycans in the interstitium and in the glycocalyx of blood vessels without commensurate water retention (sequestered sodium content [SSC]) and (3) that in patients with non-dialysis dependent chronic kidney disease, a disturbed SSC is related to capillary rarefaction and dysfunction. Therefore, the present study aims to assess the influences of both the modality (HD and HDF) and the dialysate sodium concentration (DNa) on the SSC and the MC.

Therefore the following hypotheses will be evaluated: (1, 2) treatment with hvHDF improves the SSC and MC, if compared to HD; (3, 4) disorders of the SSC and the MC are influenced by differences between the dialysate sodium [DNa] and plasma sodium [PNa] concentrations; (5) SSC and MC are interrelated in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Treatment with HD or HDF 3 x per week during at least 4 hours for at least 3 months
* Blood flow rate feasiblity of ≥350 ml/min
* Residual diuresis <200 ml/day
* Plasma Na before dialysis 137-145 mmol/L at baseline
* spKt/Vurea ≥ 1.2
* Ability to understand study procedures and willingness to provide informed consent

Exclusion Criteria:

* Severe incompliance to dialysis procedure and accompanying prescriptions, especially frequency and duration of dialysis treatment
* Life expectancy < 3 months due to non-renal disease
* Expected transplantation within 6 months
* Access recirculation > 10%
* Participation in another clinical intervention trial
* Metal implants (e.g. implantable cardioverter defibrillators)
* Severe obesity (MRI Ø 60 cm ≈ abdominal circumference ≤ 188 cm)
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Skin microcirculation | up to 20 weeks; assessed every 4 weeks before the last dialysis session of each treatment period (i.e. 5 times in total)
  Skin microcirculatory perfusion/vasoreactivity (arbitrary units) measured with a laser speckle contrast analysis (LASCA) perfusion imager
Sequestered salt content (SSC) | up to 20 weeks; assessed every 4 weeks before the last dialysis session of each treatment period (i.e. 5 times in total)
  SSC measured with a 7 Tesla 23-Sodium MRI

SECONDARY OUTCOMES:
Intradialytic hypotension | up to 4 hours (=one dialysis treatment); assessed during all dialysis sessions (12 treatments per intervention, measured 4x/hour)
  A systolic blood pressure (SBP) ≤ 90 mmHg in patients with a pre-dialysis SBP < 160 mmHg and a SBP < 100 mmHg in patients with a pre-dialysis SBP ≥ 160 mmHg.
Change in intradialytic blood pressure | up to 4 hours (=one dialysis treatment); assessed during all dialysis sessions (12 treatments per intervention, measured 4x/hour)
  Change in systolic and diastolic blood pressure (mmHg) during one dialysis session
Peridialytic blood pressure | up to 24 hours (=one interdialytic day): measured 3x/day every 4 weeks during the last interdialytic day of each treatment period (i.e. 5 times in total)
  Change in systolic and diastolic blood pressure (mmHg) between dialysis sessions
Change in CK-MB | up to 4 hours (=one dialysis treatment); measured before and immediately after the last dialysis session of each treatment period (i.e. 10 times in total)
  Marker of cardiac damage, assessment in blood from arterial line of extracorporeal circuit
Change in high sensitivity C-reactive protein (hs-CRP) | up to 4 hours (=one dialysis treatment); measured before and immediately after the last dialysis session of each treatment period (i.e. 10 times in total)
  Marker of inflammation, assessment in blood from arterial line of extracorporeal circuit
Change in interleukin-6 receptor (IL-6R) | up to 4 hours (=one dialysis treatment); measured before and immediately after the last dialysis session of each treatment period (i.e. 10 times in total)
  Marker of inflammation, assessment in blood from arterial line of extracorporeal circuit
Change in soluble CD163 (sCD163) | up to 4 hours (=one dialysis treatment); measured before and immediately after the last dialysis session of each treatment period (i.e. 10 times in total)
  Marker of inflammation, assessment in blood from arterial line of extracorporeal circuit
Change in soluble intercellular adhesion molecule-1 (s-ICAM-1) | up to 4 hours (=one dialysis treatment); measured before and immediately after the last dialysis session of each treatment period (i.e. 10 times in total)
  Marker of inflammation, assessment in blood from arterial line of extracorporeal circuit
Change in serum glycosaminoglycans | up to 4 hours (=one dialysis treatment); measured before and immediately after the last dialysis session of each treatment period (i.e. 10 times in total)
  Marker related to sequestered sodium content, assessment in blood from arterial line of extracorporeal circuit
Change in syndecan-1 | up to 4 hours (=one dialysis treatment); measured before and immediately after the last dialysis session of each treatment period (i.e. 10 times in total)
  Marker related to sequestered sodium content, assessment in blood from arterial line of extracorporeal circuit
Change in vascular endothelial growth factor C (VEGF-C) | up to 4 hours (=one dialysis treatment); measured before and immediately after the last dialysis session of each treatment period (i.e. 10 times in total)
  Marker related to sequestered sodium content, assessment in blood from arterial line of extracorporeal circuit
Change in extracellular vesicles (EVs) | up to 4 hours (=one dialysis treatment); measured before and immediately after the last dialysis session of each treatment period (i.e. 10 times in total)
  Marker for tissue-injury and inflammation, assessment in blood from arterial line of extracorporeal circuit
Change in skin microcirculation | up to 4 hours (=one dialysis treatment); measured before and immediately after the last dialysis session of each treatment period (i.e. 10 times in total)
  Change in skin microcirculatory perfusion/vasoreactivity (arbitrary units) measured with a laser speckle contrast analysis (LASCA) perfusion imager during one dialysis session. This will be assessed in 5 patients only.
Change in sequestered salt content (SSC) | up to 4 hours (=one dialysis treatment); measured before and immediately after the last dialysis session of each treatment period (i.e. 10 times in total)
  Change in SSC measured with a 7 Tesla 23-Sodium MRI during one dialysis session. This will be assessed in 5 patients only.
modified Dialysis symptom index (mDSI) | up to 20 weeks; evaluated every 4 weeks, during/after the last dialysis session of each treatment period
  Standardized questionnaire for the evaluation of physical symptoms and recovery time in dialysis patients, consisting of 13 items. Participants rate the severity of each item on a 5-point likert scale, ranging from 0 ('not at all') to 4 ('very much'). Higher scores indicate a greater perceived severity of symptoms.
Thirst distress scale (TDS) | up to 20 weeks; evaluated every 4 weeks, during/after the last dialysis session of each treatment period
  The thirst distress scale is a 6-item questionnaire that measures thirst distress on a scale from 1 to 5, where 1 corresponds to 'Strongly disagree' and 5 to 'Strongly agree'. Higher scores indicate greater perceived thirst distress.
EQ Visual analogue scale (EQ VAS) | up to 20 weeks; evaluated every 4 weeks, during/after the last dialysis session of each treatment period
  The EQ VAS records the patients's self-rated health-related quality of life on a vertical visual analogue scale where 0 means 'the worst health you can imagine' and 100 means 'the best health you can imagine'. Higher scores indicate a better perceived health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Muriel PC Grooteman, MD PhD, Principal Investigator — Amsterdam UMC

IPD SHARING:
Plan to Share IPD: No